CLINICAL TRIAL: NCT05379712
Title: A Randomized Open Label Trial of Multimodal Oral Nutritional Supplementation Versus Standard Care, to Prevent / Attenuate Malnutrition in Patients with Cancers of the Head and Neck Receiving (chemo)-radiotherapy Treatment.
Brief Title: Nutritional Supplementation in Head and Neck Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0024
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-10

CONDITIONS: Malnourishment; Nutritional Deficiency; Undernutrition
Keywords: Nutritional Support; Oral Nutritional Supplements
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized (multimodal oral nutrition therapy versus standard care), open label, parallel assignment, during cancer treatment (Baseline - Week 7 for Primary endpoint). Starting at Week 8, all patients receive the intervention arm until study ends at Week 14. Patients in the intervention arm continue the intervention, patients on the standard care arm cross over to the intervention (deferred nutrition intervention).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Nutrition Therapy (Experimental): To assess a multimodal nutrition therapy (primary nutrition intervention+ adjuvant nutrition therapy) with features adapted for patients with cancers of the head and neck receiving chemo-radiotherapy treatment, to maintain oral dietary intake during treatment. The regimen consists of 2 medical foods, each taken on an unrestricted basis (as and when preferred by each patient).
  Resource® Support Plus, a nutritionally complete Medical Food specifically for the dietary management of oncology patients with (risk of) malnutrition.
  BOOST® Soothe, a Medical Food formulated as a clear oral nutritional supplement for cancer patients with sensory alterations or oral discomfort due to cancer treatments, in particular chemo- and/or radiotherapy.
  Interventions: Other: Resource® Support Plus
- Standard of Care (No Intervention): In this setting patients rely on oral dietary intake. Ordinary, commercially available ingredients and food products are consumed. The standard of care includes weekly consultation with specialist oncology Registered Dietitian.

INTERVENTIONS:
Other: Resource® Support Plus — Nestlé Resource Support Plus® is a high energy- and protein-density Medical Food enriched with omega 3 polyunsaturated fatty acids. This is a nutritionally complete formula, in an easy to swallow, palatable, concentrated low volume, available in 2 flavours optimized for cancer patients undergoing chemotherapy and/or radiation in taste tests. It provides in a 125 mL serving: 250 kcal, 11.5 g protein and 0.95g of omega-3 fatty acid (eicosapentaenoic acid, EPA).
  Arms: Multimodal Nutrition Therapy

SUMMARY:
The purpose of this study is to determine whether multimodal nutrition therapy (primary nutrition intervention + adjuvant nutrition therapy) will support patients to optimize their total caloric intake during cancer treatment by measuring the difference in mean cumulative energy intake between the intervention and control group over the duration of cancer treatment.

DETAILED DESCRIPTION:
This will be an randomized, open label, parallel assignment study during cancer treatment (Baseline - Week 7 for Primary endpoint) comparing multimodal oral nutrition therapy versus standard care. Starting at Week 8, all patients receive the intervention arm until study ends at Week 14. Patients in the intervention arm continue the intervention, patients on the standard care arm cross over to the intervention (deferred nutrition intervention).

The primary objective is to assess a multimodal nutrition therapy with two Medical Foods (primary nutrition intervention+ adjuvant nutrition therapy) with features adapted for patients with cancers of the head and neck receiving chemo-radiotherapy treatment, to maintain oral dietary intake during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to read, understand, and sign an informed consent and must be willing to comply with study treatment and follow-up.
2. Male or female
3. ≥18 years of age
4. Histopathologically confirmed primary squamous cell carcinoma of the oral cavity and oropharynx, larynx or hypopharynx, who have agreed to receive radical intent radiotherapy as primary treatment or adjuvant treatment post-surgery, with or without platinum chemotherapy
5. Capable of volitional oral nutritional intake at baseline.
6. A diagnostic CT image taken with a maximum of 30 days before initiation of radical intent radiotherapy. If the CT scan history in the patient's clinical record does not include a study within this window, a baseline non-contrast enhanced CT abdomen will be conducted.
7. An Eastern Cooperative Oncology Group Performance Status of ≤ 2

Exclusion Criteria:

1. Fed by nasogastric tube, gastrostomy or total parenteral nutrition
2. Cancer of the nasopharynx, thyroid or salivary gland
3. Life expectancy <6 months.
4. A known hypersensitivity / allergy to the investigational product or to any ingredient in their formulations (e.g. Milk/Lactose, Fish).
5. Enrolment in any other clinical protocol or investigational study with an interventional agent or assessments that may interfere with study procedures.
6. Patients with untreated brain metastases (patients with previously resected and/or radiated brain metastases without neurologic symptoms are permitted).
7. Poorly controlled chronic illnesses or other inflammatory diseases (e.g. COPD, uncontrolled non-insulin dependent diabetes, rheumatoid arthritis).
8. In the investigators' opinion, patients who have medical conditions that could interfere with nutrient metabolism or absorption (e.g., short bowel syndrome, Crohn's disease, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in mean cumulative energy intake | Up to 14 weeks
  Energy intake is calculated from a one-day diet record in which the patient lists the identity and quantity of all foods and beverages consumed in the designated 24 hour time period at the end of each week (Baseline - Week 14).

SECONDARY OUTCOMES:
Change in mean cumulative protein take | Up to 14 Weeks
  Energy intake is calculated from a one-day diet record in which the patient lists the identity and quantity of all foods and beverages consumed in the designated 24 hour time period at the end of each week (Baseline - Week 14)
Change in body weight (kg) | Baseline-Week 14
  Change in weight (kg) from the previous week.
Change in Nutritional blood biomarkers | Baseline measures will be compared to levels at weeks 7 and 14
  A sample of blood will be collected for albumin, absolute neutrophil count, lymphocyte count, C-reactive protein, standard complete blood count-differential White Blood cell count and to measure serum CRP and albumin
Head and Neck Symptom Checklist | Up to 14 weeks
  A survey tool for HNC patient self-assessment of the presence and degree of interference with eating, over the past 3 days, of 17 symptoms known to impact dietary intake. Scores range from 34 to 170 pts, where higher scores reflect a greater presence and interference with eating. Completed at weeks 0, 4, 7, 11, 14
Taste and smell survey | Up to 14 weeks
  A survey tool for patient self-assessment of the presence, characterization and severity of taste and smell alterations. This tool yields a 'chemosensory complaint score' of up to 16 (greatest severity of taste and smell alterations). Completed at weeks 0, 4, 7, 11, 14.
Medication use for pain | Up to 14 weeks
  Use of pain medication will be captured weekly by a one- day pain medication log.
Percent oral intake from oral nutritional supplements | Up to 14 weeks
  The volume (mL) of study products consumed will be determined from the weekly one-day diet record.
Product Sensory Assessment questionnaire | Up to 14 weeks
  A product evaluation form for the Medical Nutrition products will be used to evaluate product overall sensory assessment, including acceptance and perception of characteristic product attributes that influence overall sensory acceptance. Medical Nutrition sensory acceptance will be evaluated by "overall liking" on the 9-point hedonic scale (1= dislike extremely; 9 = like extremely). Completed at weeks 0, 2, 4, 6, 8, 10, 12, 14.
Functional Assessment of Anorexia-Cachexia Treatment (FAACT) 5 Question Anorexia/Cachexia subscale (AC/S) | Up to 14 weeks
  The FAACT is a validated Quality of Life Scale to capture patient experience of cancer related cachexia - anorexia. Completed at weeks 0, 4, 7,11, 14
Cumulative energy intake (kcal/kg BW) | Up to 14 weeks
  Energy intake is calculated from a one-day diet record in which the patient lists the identity and quantity of all foods and beverages consumed in the designated 24 hour time period at the end of each week (Baseline - Week 14)
Cumulative protein take (g pro/kg BW) | Up to 14 weeks
  Protein intake is calculated from a one-day diet record in which the patient lists the identity and quantity of all foods and beverages consumed in the designated 24 hour time period at the end of each week (Baseline - Week 14)
Change in computed-tomography (CT) defined skeletal muscle and fat mass) | Within 30 days prior to start of treatment, Week 14
  Imaging for body composition (muscle, fat)
Tertiary hospital admission | Up to 14 weeks
  Review of patient medical records for instances of hospitalization with date(s) of admission falling between baseline and week 14 of study.

CONTACTS AND LOCATIONS:
Overall Officials: Vickie Baracos, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No